CLINICAL TRIAL: NCT03418064
Title: Performance of Toric Silicone Hydrogel Contact Lenses Following One Month of Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-90
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- fanfilcon A toric (Experimental): Subjects who wore fanfilcon A toric contact lens, either as the first or second lens in this cross-over study.
  Interventions: Device: Fanfilcon A toric lens
- lotrafilcon B (Active Comparator): Subjects who wore lotrafilcon B toric contact lens, either as the first or second lens in this cross-over study.
  Interventions: Device: Lotrafilcon B toric lens

INTERVENTIONS:
Device: Fanfilcon A toric lens — Contact lens
  Other Names: Avaira Vitality toric lens
  Arms: fanfilcon A toric
Device: Lotrafilcon B toric lens — Contact lens
  Other Names: AIR OPTIX for Astigmatism
  Arms: lotrafilcon B

SUMMARY:
The aim of this prospective study is to evaluate the clinical performance of fanfilcon A toric and lotrafilcon B toric contact lenses after 1 month of wear in each pair.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate the clinical performance of Avaira Vitality toric (fanfilcon A) and AIR OPTIX for Astigmatism (lotrafilcon B) contact lenses after 1 month of wear in each pair.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a contact lens spherical prescription between +6.00 to - 9.00 (inclusive)
* Have no less than -0.75D of astigmatism and no more than -2.25 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Fanfilcon A Toric, Then Lotrafilcon B Toric: Subjects wore fanfilcon A toric contact lens for 1 month, then lotrafilcon B toric contact lens.
  Fanfilcon A toric: contact lens Lotrafilcon B toric: contact lens
- Lotrafilcon B Toric, Then Fanfilcon A Toric: Subjects wore lotrafilcon B toric contact lens for 1 month, then fanfilcon A toric contact lens.
  Lotrafilcon B toric: Contact lens Fanfilcon A toric: contact lens
Period: First Intervention (1 Month)
Arm/Group | Fanfilcon A Toric, Then Lotrafilcon B Toric | Lotrafilcon B Toric, Then Fanfilcon A Toric
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Second Intervention (1 Month)
Arm/Group | Fanfilcon A Toric, Then Lotrafilcon B Toric | Lotrafilcon B Toric, Then Fanfilcon A Toric
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fanfilcon A Toric vs. Lotrafilcon B Toric Contact Lens: Each subject is randomized to wear either the fanfilcon A toric or lotrafilcon B toric contact lens as a matched pair and crossed over to second matched pair.
Arm/Group | Fanfilcon A Toric vs. Lotrafilcon B Toric Contact Lens
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 42
Region of Enrollment [Number; unit: participants]
  Mexico | 42

OUTCOME MEASURES:

1. Primary Outcome: Lens Centration
Description: Centration of lens on eye in primary gaze (1-3 scale; 1=optimal centration, 2=Decentration acceptable, slightly, 3 = decentration unacceptable)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Habitual Toric Lens at Baseline: Subjects were evaluated at baseline with their habitual toric lenses.
Arm/Group | Habitual Toric Lens at Baseline
Number analyzed (Participants) | 42
Participants
  1-Optimal Centration | 41
  2-Decentration acceptable | 1
  3-Decentranation Unacceptable | 0

2. Primary Outcome: Lens Centration
Description: as for outcome 1
Time Frame: Dispense
Measure: Count of Participants; unit: Participants
Groups:
- Fanfilcon A Toric at Dispense: Subjects who wore fanfilcon A toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Fanfilcon A toric lens: Contact lens
- Lotrafilcon B Toric at Dispense: Subjects who wore lotrafilcon B toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Lotrafilcon B toric lens: Contact lens
Arm/Group | Fanfilcon A Toric at Dispense | Lotrafilcon B Toric at Dispense
Number analyzed (Participants) | 42 | 42
Participants
  1-Optimal Centration | 42 | 42
  2-Decentration acceptable | 0 | 0
  3-Decentranation Unacceptable | 0 | 0

3. Primary Outcome: Lens Centration
Description: as for outcome 1
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Groups:
- Fanfilcon A Toric Lens at 1 Month: Subjects who wore fanfilcon A toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Fanfilcon A toric lens: Contact lens
- Lotrafilcon B Toric at 1 Month: Subjects who wore lotrafilcon B toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Lotrafilcon B toric lens: Contact lens
Arm/Group | Fanfilcon A Toric Lens at 1 Month | Lotrafilcon B Toric at 1 Month
Number analyzed (Participants) | 42 | 42
Participants
  1-Optimal Centration | 42 | 42
  2-Decentration acceptable | 0 | 0
  3-Decentranation Unacceptable | 0 | 0

4. Primary Outcome: Corneal Coverage
Description: Evaluate corneal coverage of contact lens (Yes=Full, No=Incomplete)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Habitual Toric Lens at Baseline
Number analyzed (Participants) | 42
Participants
  Full Coverage (Yes) | 42
  Incomplete (No) | 0

5. Primary Outcome: Corneal Coverage
Description: Evaluate corneal coverage of contact lens (Yes=Full, No=Incomplete)
Time Frame: Dispense
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A Toric at Dispense | Lotrafilcon B Toric at Dispense
Number analyzed (Participants) | 42 | 42
Participants
  Full Coverage (Yes) | 42 | 42
  Incomplete (No) | 0 | 0

6. Primary Outcome: Corneal Coverage
Description: Evaluate corneal coverage of contact lens (Yes=Full, No=Incomplete)
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A Toric Lens at 1 Month | Lotrafilcon B Toric at 1 Month
Number analyzed (Participants) | 42 | 42
Participants
  Full Coverage (Yes) | 42 | 42
  Incomplete (No) | 0 | 0

7. Primary Outcome: Post-blink Movement
Description: Amount of lens movement after blink (0-4 scale, 0=insufficient, unacceptable movement, 2=optimal movement, 3=moderate, but acceptable movement 4=excessive, unacceptable movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Habitual Toric Lens at Baseline
Number analyzed (Participants) | 42
score on a scale | 2.17 (0.5)

8. Primary Outcome: Post-blink Movement
Description: as for outcome 7
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fanfilcon A Toric at Dispense | Lotrafilcon B Toric at Dispense
Number analyzed (Participants) | 42 | 42
score on a scale | 2.02 (0.2) | 2.05 (0.5)

9. Primary Outcome: Post-blink Movement
Description: as for outcome 7
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fanfilcon A Toric Lens at 1 Month | Lotrafilcon B Toric at 1 Month
Number analyzed (Participants) | 42 | 42
score on a scale | 2.00 (0.0) | 2.10 (0.4)

10. Primary Outcome: Overall Fit Acceptance
Description: Assessed by investigator based on lens fit alone (0-4 scale; 0=should not be worn, 4=perfect)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A Toric Contact Lens Dispense: Subjects who wore fanfilcon A toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Fanfilcon A toric lens: Contact lens
- Lotrafilcon B Toric Contact Lens Dispense: Subjects who wore lotrafilcon B toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  lotrafilcon B toric lens: Contact lens
Arm/Group | Fanfilcon A Toric Contact Lens Dispense | Lotrafilcon B Toric Contact Lens Dispense
Number analyzed (Participants) | 42 | 42
units on a scale | 3.8 (0.5) | 2.4 (1.0)

11. Primary Outcome: Overall Fit Acceptance
Description: Assessed by investigator based on lens fit alone (0-4 scale; 0=should not be worn, 4=perfect)
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A Toric Contact Lens 1 Month: Subjects who wore fanfilcon A toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  Fanfilcon A toric lens: Contact lens
- Lotrafilcon B Toric Contact Lens 1 Month: Subjects who wore lotrafilcon B toric contact lens for 1 month, either randomized as the first or second lens in this cross-over study.
  lotrafilcon B toric lens: Contact lens
Arm/Group | Fanfilcon A Toric Contact Lens 1 Month | Lotrafilcon B Toric Contact Lens 1 Month
Number analyzed (Participants) | 42 | 42
units on a scale | 3.9 (0.4) | 2.5 (0.9)

12. Secondary Outcome: Average Hours of Wear Per Day
Description: Number of hours lenses are worn per day
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours per day
Groups:
- Habitual Toric Lens: Subjects were evaluated at baseline with their habitual toric lenses.
Arm/Group | Habitual Toric Lens
Number analyzed (Participants) | 42
hours per day | 13.8 (3.0)

13. Secondary Outcome: Average Hours of Wear Per Day
Description: Number of hours lenses are worn per day
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Fanfilcon A Toric Lens at 1 Month | Lotrafilcon B Toric at 1 Month
Number analyzed (Participants) | 42 | 42
hours per day | 14.1 (2.9) | 14.0 (2.6)

14. Secondary Outcome: Average Comfortable Wearing Time
Description: Typical time of day when subject first experiences lens awareness or irritation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Habitual Toric Lens
Number analyzed (Participants) | 42
hours per day | 11.5 (2.9)

15. Secondary Outcome: Average Comfortable Wearing Time
Description: Typical time of day when subject first experiences lens awareness or irritation
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Fanfilcon A Toric Lens at 1 Month | Lotrafilcon B Toric at 1 Month
Number analyzed (Participants) | 42 | 42
hours per day | 11.4 (3.3) | 11.0 (3.4)

ADVERSE EVENTS:
Time Frame: From dispense to completion of follow up, up to 1 month.
Groups:
- Lotrafilcon B Toric: Subjects who wore lotrafilcon B toric contact lens, either as the first or second lens in this cross-over study.
  Lotrafilcon B toric lens: Contact lens
Arm/Group | Fanfilcon A Toric | Lotrafilcon B Toric
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator cannot publish / present data without prior consent from CooperVision.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03418064/Prot_SAP_000.pdf